CLINICAL TRIAL: NCT06505499
Title: Gait Profile Score in Children With Cerebral Palsy (CP): Influence of the CP Type, Treatment With Botulinum Injection and Multilevel Surgery
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: IRBN402024/CHUSTE
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy; Gait Disorders in Children
Keywords: Cerebral palsy; Gait profile score; Botulinum toxin injection; Multilevel surgery
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EXPERIMENTAL GROUP: Children and teenagers with CP with an instrumented gait analysis performed since 2019.
  Interventions: Other: Gait Profile Score; Other: Gait Visual Score

INTERVENTIONS:
Other: Gait Profile Score — Gait Profile Score in degrees, calculated from kinematic raw data with the Gdi_GPS_calculator spreadsheet developed by Baker (2009).
Other: Gait Visual Score — Gait Visual Score in degrees, calculated from kinematic raw data with the Gdi_GPS_calculator spreadsheet developed by Baker (2009)

SUMMARY:
Instrumented three dimensional gait analysis (3DGA) permits to record spatial, temporal, kinetics, kinematics and electromyographic (EMG) parameters in order to understand gait impairment in children and teenagers with cerebral palsy (CP). Nowadays, single-event multilevel surgery in subjects with CP cannot be performed without 3DGA. However, interpretation of multiple and interdependent data remains complex for the clinician. To address this issue, gait statistical index have been developed to give a single measure of the quality of the gait pattern. Among actual index, the Gait Profile Score (GPS), developed by Baker et al (2009), measure the deviation of kinematics parameters from a controlled dataset. The GPS can be divided in nine Gait Variable Score (GVS), corresponding to major lower limb joints: the MAP (Movement Analysis Profile). Many studies have reported the interest of the GPS to analysis gait of subjects with CP: good inter-session reliability, predictor of postoperative kinematic improvement, minimal clinical threshold calculated at 1.6°, significant relationship with clinical data (joint contractures), and sensibility to change after a single-event multilevel surgery.

ELIGIBILITY:
Inclusion Criteria:

* Etiology of cerebral palsy
* Unilateral, bilateral, triplegic or quadriplegic forms of cerebral palsy.
* 6 to 18 years old
* GMFCS (Gross Motor Function Classification System) I to III
* Instrumented gait analysis of the laboratory of St-Etienne
* Absence of botulinum toxin injection or serial casting in the three months after a first instrumented gait analysis.

Exclusion Criteria:

* Etiology others than cerebral palsy as defined classically (ex: ischemic infarcts in a child older than two years).
* Previous surgery in lower-limb.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children and adolescents with cerebral palsy treated at the Saint-Etienne University Hospital will be included.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Degrees of Gait Profile Score overall | Day 1
  Analyze Degrees of Gait Profile Score overall

SECONDARY OUTCOMES:
Gait Profile Score right | Month 2
  Analyze Gait Profile Score right.
Gait Profile Score left | Year 2
  Analyze Gait Profile Score left.

CONTACTS AND LOCATIONS:
Overall Officials: Clément BOULARD, physiotherapist, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- Chu de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No